CLINICAL TRIAL: NCT03299790
Title: Effect of High-intensity Interval Training on Cardiac Function and Regulation of Glycemic Control in Diabetic Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Dominique Hansen, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HITDCM01
Record Dates: First submitted 2017-09-12; First posted 2017-10-03 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Cardiomyopathies; Type2 Diabetes
Keywords: Type 2 diabetes; Diabetic cardiomyopathy; Cardiac function; Exercise echocardiography; Exercise training
MeSH Terms: conditions — Diabetic Cardiomyopathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- training group 1: HIIT (Active Comparator): high-intensity interval exercise training group (T2DM patients)
  Interventions: Other: high-intensity interval exercise training (HIIT)
- training group 2: MIT (Active Comparator): moderate-intensity exercise training group (T2DM patients)
  Interventions: Other: moderate-intensity exercise training (MIT)
- Detraining period (No Intervention): Follow-up: detraining of group 1 and 2 (T2DM patients)
- Healthy controls (No Intervention)

INTERVENTIONS:
Other: high-intensity interval exercise training (HIIT) — This program includes 24 weeks of exercise training and is divided in different phases (phase 1: week 1-2, equal to the MIT group, phase 2: week 3-6, 6 bouts of high-intensity exercise, phase 3: week 7-12, 7 bouts of high-intensity exercise, phase 4: week 13-24, 8 bouts of high-intensity exercise). The exercise training program consists of 3 exercise sessions per week (for 6 months).
  Arms: training group 1: HIIT
Other: moderate-intensity exercise training (MIT) — This program includes 24 weeks of exercise training and is not devided in phases. The exercise training program consists of 3 endurance exercise sessions per week (for 6 months). The total exercise volume equals the exercise volume of the HIIT group.
  Arms: training group 2: MIT

SUMMARY:
According to data of the International Diabetes Federation (IDF), diabetes in general affects approximately 415 million people worldwide and this number is still increasing. Cardiovascular diseases, one of the major complications of diabetes, are the leading cause of mortality and morbidity in the diabetic population. One of the cardiovascular complications is diabetic cardiomyopathy, in which structural and functional changes occur in the heart impairing cardiac function.

Exercise training has already proven the benefits on glycemic control in diabetes. This is also the case for the effects on cardiac function. However, as results are conflicting, it remains unclear which elements of exercise training should be focused on. For instance, high-intensity interval training (HIIT) is gaining interest as positive effects are already shown on glycemic control. Therefore, the potential of HIIT to improve cardiac function in diabetes should be investigated. Further on, the effects of exercise training on cardiac function are mainly investigated during rest by the use of transthoracic echocardiography. Therefore, as data are lacking, it remains unclear how the diabetic heart functions during exercise.

The aim of the present study is to investigate the effects of different training modalities (e.g. HIIT) on heart function in diabetes both during rest and during exercise itself. Therefore, cardiac function will be evaluated by the use transthoracic (exercise) echocardiography. This will be combined by the evaluation of several biochemical parameters.

The results will provide more insight in the pathology of diabetic cardiomyopathy as well as the potential of exercise training for this cardiovascular complication. Eventually, this research will contribute to the optimization of exercise programs for patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patients:

  * BMI > 20kg/m²
  * diagnosis of T2DM as stated in guidelines of ADA (American Diabetes Association)
  * stable medication for at least 3 months
* Healthy controls:

  * BMI > 20kg/m²
  * no diabetes

Exclusion Criteria:

* iron deficiency anemia
* participation in another clinical trial
* heart diseases: CAD (coronary artery disease), ischemia, valvular diseases, congenital heart diseases
* neurological, pneumological, oncological, orthopedic disorders
* diabetes complications: renal diseases, retinopathy

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Transthoracic echocardiography (TTE) during excercise | day 1
  heart function during exercise by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) during excercise | month 3
  heart function during exercise by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) during excercise | month 6
  heart function during exercise by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) during excercise | month 12
  heart function during exercise by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) | day 1
  heart function in rest by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) | month 3
  heart function in rest by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) | month 6
  heart function in rest by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
Transthoracic echocardiography (TTE) | month 12
  heart function in rest by means of standard echocardiography: evaluation of diastolic and systolic function (mitral inflow pattern, ejection fraction, tissue doppler imaging, strain rate analyses,…) and cardiac structure (left ventricle mass, intraventricular wall mass,…)
ECG (Electrocardiogram) during excercise | month 3
  ECG during excercise (an incremental exercise test on a cycle)
ECG (Electrocardiogram) during excercise | month 12
  ECG during excercise (an incremental exercise test on a cycle)
ECG (Electrocardiogram) | month 3
  ECG in rest
ECG (Electrocardiogram) | month 12
  ECG in rest

SECONDARY OUTCOMES:
Glycemic control | day 1
  glycemic concentrations, HbA1c levels, insulin sensitivity, inflammation, cardiac biomarkers
Glycemic control | month 3
  glycemic control, insulin sensitivity, inflammation, cardiac biomarkers
Glycemic control | month 6
  glycemic concentrations, HbA1c levels, insulin sensitivity, inflammation, cardiac biomarkers
Glycemic control | month 12
  glycemic concentrations, HbA1c levels, insulin sensitivity, inflammation, cardiac biomarkers
Insulin metabolism | day 1
  Fasting serum insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test (75g)
Insulin metabolism | month 3
  Fasting serum insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test (75g)
Insulin metabolism | month 6
  Fasting serum insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test (75g)
Insulin metabolism | month 12
  Fasting serum insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test (75g)
Cardiac function | day 1
  Cardiac biomarkers (brain-derived natriuretic peptide (BNP) levels, cardiac troponin levels)
Cardiac function | month 3
  Cardiac biomarkers (BNP levels, cardiac troponin levels)
Cardiac function | month 6
  Cardiac biomarkers (BNP levels, cardiac troponin levels)
Cardiac function | month 12
  Cardiac biomarkers (BNP levels, cardiac troponin levels)
Inflammation and oxidative stress | day 1
  C reactive protein (CRP) levels, tumor necrosis factor-(TNF)alpha levels, interleukin (IL)-10 (interleukin) levels, oxidative stress markers (superoxide dismutase (SOD), malondialdehyde (MDA), glutathione peroxidase (GPX))
Inflammation and oxidative stress | month 3
  CRP levels, TNF-alpha levels, IL-10 levels, oxidative stress markers (SOD, MDA, GPX)
Inflammation and oxidative stress | month 6
  CRP levels, TNF-alpha levels, IL-10 levels, oxidative stress markers (SOD, MDA , GPX)
Inflammation and oxidative stress | month 12
  CRP levels, TNF-alpha levels, IL-10 levels, oxidative stress markers (SOD, MDA, GPX)
body composition | day 1
  body composition, measured using dual x-ray absorptiometry
body composition | month 6
  body composition, measured using dual x-ray absorptiometry
Maximal oxygen uptake (ml/O2/kg/min) | day 1
  exercise capacity measured using indirect calorimetry and an incremental bicycle exercise protocol
Maximal oxygen uptake (ml/O2/kg/min) | month 3
  exercise capacity measured using indirect calorimetry and an incremental bicycle exercise protocol
Maximal oxygen uptake (ml/O2/kg/min) | month 6
  exercise capacity measured using indirect calorimetry and an incremental bicycle exercise protocol
Maximal oxygen uptake (ml/O2/kg/min) | month 12
  exercise capacity measured using indirect calorimetry and an incremental bicycle exercise protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

REFERENCES:
- [Derived] Van Ryckeghem L, Keytsman C, De Brandt J, Verboven K, Verbaanderd E, Marinus N, Franssen WMA, Frederix I, Bakelants E, Petit T, Jogani S, Stroobants S, Dendale P, Bito V, Verwerft J, Hansen D. Impact of continuous vs. interval training on oxygen extraction and cardiac function during exercise in type 2 diabetes mellitus. Eur J Appl Physiol. 2022 Apr;122(4):875-887. doi: 10.1007/s00421-022-04884-9. Epub 2022 Jan 17. PMID 35038022
- [Derived] Van Ryckeghem L, Keytsman C, Verboven K, Verbaanderd E, Frederix I, Bakelants E, Petit T, Jogani S, Stroobants S, Dendale P, Bito V, Verwerft J, Hansen D. Exercise capacity is related to attenuated responses in oxygen extraction and left ventricular longitudinal strain in asymptomatic type 2 diabetes patients. Eur J Prev Cardiol. 2022 Jan 11;28(16):1756-1766. doi: 10.1093/eurjpc/zwaa007. PMID 33623980
- [Derived] Van Ryckeghem L, Keytsman C, Verbaanderd E, Frederix I, Bakelants E, Petit T, Jogani S, Stroobants S, Dendale P, Bito V, Verwerft J, Hansen D. Asymptomatic type 2 diabetes mellitus display a reduced myocardial deformation but adequate response during exercise. Eur J Appl Physiol. 2021 Mar;121(3):929-940. doi: 10.1007/s00421-020-04557-5. Epub 2021 Jan 8. PMID 33417036